CLINICAL TRIAL: NCT04621708
Title: Pilot Study of the Safety and Tolerability of Left Dorsolateral Prefrontal Cortex Intermittent Theta Burst rTMS for Major Depressive Disorder in Multiple Sclerosis
Brief Title: Pilot Study of the Safety and Tolerability of L-DLPFC iTBS rTMS for MDD in MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Peter Giacobbe, Clinical Head, Harquail Centre for Neuromodulation, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1563
Record Dates: First submitted 2020-10-21; First posted 2020-11-09 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis; Major Depressive Disorder
Keywords: MS; MDD
MeSH Terms: conditions — Multiple Sclerosis; Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This study is designed as an open-label pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Left DLPFC iTBS rTMS (Experimental)
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Left DLPFC iTBS rTMS

SUMMARY:
The main purpose of this study is to investigate the safety and tolerability of intermittent Theta Burst (iTBS) repetitive transcranial magnetic stimulation (rTMS), its effectiveness in alleviating depressive symptoms as well as its effects on cognition. Although iTBS rTMS is approved for use, there have been no safety and tolerability evaluations of this form of rTMS in Multiple Sclerosis (MS).

DETAILED DESCRIPTION:
The main purpose of this study is to investigate the safety and tolerability of intermittent Theta Burst (iTBS), its effectiveness in alleviating depressive symptoms, concomitant neuropsychiatric symptoms such as anxiety and fatigue in people with MS, as well as its effects on cognition. Although iTBS repetitive transcranial magnetic stimulation (rTMS) is approved for use in major depressive disorder (MDD), there have been no safety and tolerability evaluations of this form of rTMS in Multiple Sclerosis (MS) patient with MDD. Although iTBS rTMS has previously been found safe and effective for treating spasticity in people with MS, this will be the first study to investigate the safety and tolerability of Left Dorsolateral Prefrontal Cortex (L-DLPFC) iTBS rTMS for MDD in MS

This study is designed as an open-label pilot study. Participants will undergo baseline evaluations to confirm a diagnosis of MDD and to assess your eligibility for rTMS treatment. If deemed eligible, participants will receive iTBS treatment. iTBS is a form of rTMS approved by Health Canada for treatment of MDD. iTBS rTMS treatment involves 3 minutes of non-invasive brain stimulation, 5 days a week, for 4 weeks, for a total of 20 treatments. While receiving iTBS rTMS, participants will be seen daily by the rTMS operator who is a mental health nurse. While receiving iTBS rTMS, participants will see the research coordinator and study psychiatrist on a weekly basis, to complete clinical assessments to evaluate their neuropsychiatric symptoms and assess any side effects from the rTMS procedure. As part of the suggested pathophysiological profile of depression the levels of inflammatory cytokines tumor necrosis factor ⍺ (TNF-⍺) and interleukin-6 (IL-6) have shown elevated concentration levels in plasma of depressed compared to non-depressed individuals. In this study, we aim to investigate the levels of these inflammatory cytokine markers and their change with iTBS.

ELIGIBILITY:
Inclusion criteria

1. Men and women ≥18 and ≤70 years of age, inclusive.
2. History of MS confirmed by a neurologist.
3. Patients who are able and willing to give consent and able to adhere to treatment schedule and attend study visits, as determined by study psychiatrist
4. DSM-V diagnosis of Major Depressive Disorder (MDD)
5. Moderate severity with a Hamilton Depression Rating Scale (HAMD) at least 16
6. Patients have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening
7. Pass the TMS safety screening questionnaire
8. Women of childbearing potential must agree to use a barrier contraception method throughout the study.

Exclusion criteria

1. Active substance abuse or dependence in the last three months, except nicotine
2. Active suicidal intent
3. Currently pregnant (as determined by history and serum HCG) or lactating.
4. A diagnosis of Bipolar Disorder
5. A history of past or current psychotic symptoms
6. Diagnosis of obsessive-compulsive disorder, post-traumatic stress disorder (current or within the last year), assessed by a study investigator to be primary and causing greater impairment than MDD
7. Having failed a course of ECT in the current episode or previous episode
8. Previous trial of rTMS
9. Personality disorder deemed to be primary pathology
10. If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
11. Clinically significant laboratory abnormality, in the opinion of the investigator
12. Unstable medical illness
13. Contraindication to rTMS, e.g. presence of cardiac pacemaker, intracranial implant, or metal in the cranium
14. Currently on more than 2 mg of lorazepam or equivalent
15. History of seizures, or currently on anticonvulsant for seizures
16. Concurrent use of a medication that may lower the seizure threshold, in the opinion of the investigator e.g. stimulant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms | Baseline and 4 weeks post-treatment
  The primary outcome measure will be the reduction in depressive symptoms as measured by the Hamilton Depression Rating Scale-17 at the end of the 4-week trial of iTBS rTMS. This will be measured as both a continuous variable (score on HAMD-17 at week 4 - score on HAMD-17 at week 0 pre-treatment) and a categorical one (i.e. the response rates of >50% reduction from baseline HAMD-17 and remission rates defined as HAMD-17 <7).

SECONDARY OUTCOMES:
Change in anxiety and depressive symptoms | Baseline and 4 weeks post-treatment
  Change in anxiety and depressive symptoms as measured by the self-report Hospital Anxiety and Depression Scale (HADS)-17 at the end of the 4-week trial of iTBS rTMS.
Change in fatigue, severity and impact | Baseline and 4 weeks post-treatment
  Change in fatigue, severity and impact, measured by the self-report Fatigue Severity Scale (FSS)
Change in Neuropsychological function | Baseline and 4 weeks post-treatment
  Change in Neuropsychological function, measured subjectively through the Perceived Deficits Questionnaire (PDQ-5) and objectively by the SDMT and computerized CANTAB neuropsychological tasks
Change in fatigue, severity and impact | Baseline and 4 weeks post-treatment
  Change in fatigue, severity and impact, measured by the Modified Fatigue Impact Scale (MFIS), respectively
Change in Neuropsychological function | Baseline and 4 weeks post-treatment
  Change in Neuropsychological function, measured objectively by the computerized CANTAB neuropsychological tasks

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada